CLINICAL TRIAL: NCT01198002
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of LY2127399 in Patients With Moderate to Severe Rheumatoid Arthritis (RA) Who Had an Inadequate Response to Methotrexate Therapy (FLEX M)
Brief Title: A Rheumatoid Arthritis Study in Participants on a Background Treatment of Methotrexate
Acronym: FLEX M
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated not based on safety concerns, but due to insufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11352; H9B-MC-BCDM (Other: Eli Lilly and Company); CTRI/2011/07/001870 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 120 milligrams (mg) LY2127399 (Experimental): Given every 4 weeks (Q4W) for 100 weeks. Participants receive a 240 mg loading dose when initiating treatment. During the Treatment Period, for blinding purposes, participants will alternate injections of LY2127399 and injections of placebo every 2 weeks (Q2W).
  At Weeks 16 and 52, responders will receive 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 100-week treatment period.
  At Week 16, non-responders (NR) will receive 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
  Interventions: Drug: LY2127399; Drug: Placebo Q4W; Drug: Methotrexate
- 90 mg LY2127399 (Experimental): Given Q2W for 100 weeks. Participants receive a 180 mg loading dose when initiating treatment.
  At Weeks 16 and 52, responders will receive 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q4W for the rest of the 100-week treatment period.
  At Week 16, NR will receive 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
  Interventions: Drug: LY2127399; Drug: Methotrexate
- Placebo (Placebo Comparator): Given Q2W for 52 weeks. At Week 16, responders will receive 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the 52 weeks.
  At Week 52, responders are randomized to receive 1 of the 2 doses of LY2127399, with loading dose of 240 mg or 180 mg of LY2127399, followed by 120 mg of LY2127399 Q4W or 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
  At Week 16, NR will receive a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
  Interventions: Drug: LY2127399; Drug: Placebo Q2W; Drug: Methotrexate

INTERVENTIONS:
Drug: LY2127399 — Administered Subcutaneously (SC)
Drug: Placebo Q2W — Administered SC
  Arms: Placebo
Drug: Placebo Q4W — Administered SC
  Arms: 120 milligrams (mg) LY2127399
Drug: Methotrexate — Methotrexate is a background therapy.

SUMMARY:
The primary purpose of this study is to help answer if LY2127399 is safe and effective in the treatment of rheumatoid arthritis while on a background treatment of methotrexate.

This study is comprised of 3 periods:

Period 1: 52-week blinded treatment

Period 2: additional 48-week unblinded treatment

Period 3: 48-week post-treatment follow-up

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis (RA) of more than 6 months and less than 15 years
* Regular use of methotrexate (MTX) in the past 12 weeks, with the dose being stable during the past 8 weeks
* At least 8 tender and swollen joints
* At least one erosion of a hand or foot joint observed on an X-ray
* An abnormally high C-reactive protein (CRP) level or erythrocyte sedimentation rate (ESR)
* Positive for rheumatoid factor (RF) or anti-cyclic citrullinated peptide (CCP) antibody
* Woman must not be pregnant, breastfeeding, or become pregnant during the study

Exclusion Criteria:

* Use of unstable doses of non-steroidal anti-inflammatory drugs (NSAIDS) in the past 6 weeks
* Steroid injection or intravenous (iv) infusion in the last 6 weeks
* Use of more than 10 milligrams/day (mg/day) of oral steroids in the last 6 weeks
* History of an inadequate response to a biologic disease-modifying anti-rheumatic drug (DMARD)
* History of a serious reaction to other biological DMARDs
* History of the use of rituximab or other B cell therapy
* Use of DMARDS other than MTX, hydroxychloroquine, or sulfasalazine within the last 8 weeks
* Use of leflunomide within the last 12 weeks (unless cholestyramine was used to speed up the elimination of leflunomide)
* Surgery on a joint or other major surgery less than 2 months ago, or plans to have joint surgery or major surgery during the study
* Active fibromyalgia, juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, or other systemic inflammatory condition except RA
* Cervical cancer or squamous skin cancer within the past 3 years, or other cancer within the past 5 years
* Received a live vaccine received within the past 12 weeks (for example, vaccines for measles, mumps, rubella, and chicken pox, and nasal-spray flu vaccines)
* Hepatitis or human immunodeficiency virus (HIV)
* A serious bacterial infection (for example, pneumonia or cellulitis) within 3 months or a serious bone or joint infection within 6 months
* Symptoms of herpes zoster or herpes simplex within the last month
* Active or latent tuberculosis (TB)
* Current symptoms of a serious disorder or illness
* Use of an investigational drug within the last month
* History of the use of rituximab, any other B cell targeted biotherapy, or denosumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1041 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (233):
- United States (75):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paradise Valley, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hot Springs, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hemet, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boynton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeBary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinellas Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venice, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockbridge, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shawnee Mission, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bingham Farms, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sanford, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erie, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenixville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pottstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Watertown, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nassau Bay, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Richland Hills, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waco, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Racine, Wisconsin
- Argentina (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luján
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campbelltown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern East
- Brazil (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caxias do Sul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juiz de Fora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Bulgaria (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burgas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pleven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rousse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sevlievo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varna
- Colombia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bogotá
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medellín
- Croatia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Opatija
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rijeka
- Hungary (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balassagyarmat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiskunhalas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sátoraljaújhely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szikszó
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- India (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucknow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mysore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nellore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surat
- Japan (26):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Japan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ohita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipedos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- Malaysia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kota Bharu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perak
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Putrajaya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarawak
- Mexico (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrio San Mateo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Querétaro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tijuana
- New Zealand (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotorua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tauranga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timaru
- Poland (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Działdowo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Płock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Włoszczowa
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
- Russia (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnaul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kemerovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khanty-Mansiysk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petrozavodsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ryazan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Voronezh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl
- Slovakia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunajská Streda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piešťany
- South Africa (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benoni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limpopo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
- South Korea (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Sri Lanka (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colombo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalubowila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nugegoda
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keelung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Ukraine (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia

REFERENCES:
- [Derived] Smolen JS, Weinblatt ME, van der Heijde D, Rigby WF, van Vollenhoven R, Bingham CO 3rd, Veenhuizen M, Gill A, Zhao F, Komocsar WJ, Berclaz PY, Ortmann R, Lee C. Efficacy and safety of tabalumab, an anti-B-cell-activating factor monoclonal antibody, in patients with rheumatoid arthritis who had an inadequate response to methotrexate therapy: results from a phase III multicentre, randomised, double-blind study. Ann Rheum Dis. 2015 Aug;74(8):1567-70. doi: 10.1136/annrheumdis-2014-207090. Epub 2015 Apr 14. PMID 25873635

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study had a blinded Treatment Period 1 (Weeks 0-52), a non-blinded Treatment Period 2 (Weeks 52-100) and a post-treatment follow-up (24-48 weeks in length). All participants were assessed for nonresponse at Week 16 with non-responders (NR) defined as participants with <20% improvement from baseline in both tender and swollen joint counts.
Groups:
- 120 mg LY2127399: Treatment Period 1 (Weeks 0-52): A loading dose of 240 milligrams (mg) (2 injections of 120 mg) of LY2127399, followed by maintenance dosing of 120 mg of LY2127399 administered subcutaneously (SC) every 4 weeks (Q4W). For blinding purposes, participants alternated injections of LY2127399 and injections of placebo every 2 weeks (Q2W).
  At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
- 90 mg LY2127399: Treatment Period 1 (Weeks 0-52): A loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W.
  At Week 16, responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, Week 16 responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
- Placebo: Treatment Period 1 (Weeks 0-52): A loading dose of 2 injections of placebo, followed by maintenance dosing of 1 injection of placebo administered SC Q2W.
  At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, responders were randomized to receive either 2 injections of 120 mg of LY2127399, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2 or 2 injections of 90 mg of LY2127399, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
  At Week 16, NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
Period: Treatment Period 1 (Weeks 0-52)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Started | 345 | 347 | 349
Received at Least 1 Dose of Study Drug | 345 | 345 | 348
Week 16 NR | 58 | 62 | 90
Post-Treatment Follow-Up Population | 293 | 303 | 307
Completed | 70 (Those who completed 52-week Treatment Period 1 including both Week 16 responders and NR.) | 73 (Those who completed 52-week Treatment Period 1 including both Week 16 responders and NR.) | 80 (Those who completed 52-week Treatment Period 1 including both Week 16 responders and NR.)
Not Completed | 275 | 274 | 269
Not completed — Adverse Event | 18 | 11 | 11
Not completed — Death | 2 | 0 | 1
Not completed — Lack of Efficacy | 10 | 9 | 6
Not completed — Entry Criteria Not Met | 1 | 3 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 16 | 21 | 12
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Protocol Violation | 14 | 10 | 10
Not completed — Sponsor Decision | 213 | 216 | 224
Period: Treatment Period 2 (Weeks 52-100)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Started | 70 | 73 | 80
Completed | 1 | 0 | 2
Not Completed | 69 | 73 | 78
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lack of Efficacy | 3 | 1 | 1
Not completed — Entry Criteria Not Met | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Sponsor Decision | 62 | 70 | 75

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 120 mg LY2127399: Treatment Period 1 (Weeks 0-52): A loading dose of 240 mg (2 injections of 120 mg) of LY2127399, followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
- Total: Total of all reporting groups
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo | Total
Number analyzed (Participants) | 345 | 347 | 349 | 1041
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.8) | 52.8 (10.9) | 52.9 (11.5) | 53.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 291 | 292 | 877
  Male | 51 | 56 | 57 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 67 | 61 | 191
  Not Hispanic or Latino | 140 | 131 | 140 | 411
  Unknown or Not Reported | 142 | 149 | 148 | 439
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 18 | 15 | 53
  Asian | 100 | 102 | 101 | 303
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 22 | 19 | 22 | 63
  White | 191 | 197 | 200 | 588
  More than one race | 9 | 7 | 7 | 23
  Unknown or Not Reported | 3 | 3 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56 | 55 | 56 | 167
  Taiwan | 10 | 11 | 10 | 31
  Slovakia | 4 | 3 | 4 | 11
  Ukraine | 23 | 22 | 23 | 68
  Lithuania | 6 | 6 | 8 | 20
  Russia | 23 | 25 | 24 | 72
  Colombia | 19 | 21 | 11 | 51
  Sri Lanka | 1 | 2 | 2 | 5
  India | 5 | 5 | 4 | 14
  Hungary | 8 | 9 | 8 | 25
  Mexico | 20 | 16 | 28 | 64
  Argentina | 17 | 17 | 16 | 50
  Malaysia | 2 | 3 | 3 | 8
  Brazil | 14 | 14 | 13 | 41
  Poland | 33 | 34 | 33 | 100
  Croatia | 1 | 0 | 1 | 2
  Romania | 0 | 2 | 2 | 4
  South Africa | 16 | 16 | 16 | 48
  Bulgaria | 11 | 11 | 10 | 32
  Japan | 52 | 53 | 53 | 158
  New Zealand | 1 | 0 | 1 | 2
  South Korea | 23 | 22 | 23 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 20% Response (ACR20) at Week 24
Description: ACR Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis (RA). ACR20 Responder: had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and C-reactive protein (CRP). Percentage of participants achieving ACR20 response=(number of ACR20 responders) / (number of participants treated) * 100. All NR at Week 16 as well as all participants who discontinued study treatment at any time for any reason were defined as NR starting at that time-point and going forward, including Week 24 endpoint.
Time Frame: Baseline through 24 weeks
Population: All randomized participants with evaluable ACR20 responder data. If participant's CRP was missing, last post-baseline value was used. If ACR was missing after carrying forward CRP, last post-baseline ACR response was used. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Groups:
- 120 mg LY2127399: Treatment Period 1 (Weeks 0-52): A loading dose of 240 mg (2 injections of 120 mg) of LY2127399, followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2.
- 90 mg LY2127399: Treatment Period 1 (Weeks 0-52): A loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W.
  At Week 16, responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, Week 16 responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
- Placebo: Placebo Treatment Period 1 (Weeks 0-52): A loading dose of 2 injections of placebo, followed by maintenance dosing of 1 injection of placebo administered SC Q2W.
  At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, responders were randomized to receive either 2 injections of 120 mg of LY2127399, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2 or 2 injections of 90 mg of LY2127399, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 330 | 332 | 335
percentage of participants | 29.7 | 32.8 | 25.1

2. Primary Outcome: Change From Baseline to Week 52 in Van Der Heijde Modified Total Sharp Score (mTSS)
Description: The mTSS quantifies the extent of bone erosions and joint space narrowing for 44 and 42 joints. X-rays of the hands/wrists and feet are scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosions scores (range = 0 to 220 for 44 joints) and narrowing scores (range = 0 to 168 for 42 joints) were added to obtain the mTSS (range = 0 [normal] to 388 [maximal disease]). Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 52 Weeks
Population: All randomized participants with evaluable mTSS data. A linear extrapolation method was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo Treatment Period 1 (Weeks 0-52): A loading dose of 2 injections of placebo, followed by maintenance dosing of 1 injection of placebo administered SC Q2W.
  At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, responders were randomized to receive either 2 injections of 120 mg of LY2127399, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2 or 2 injections of 90 mg of LY2127399, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
  At Week 16, NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 295 | 304 | 306
units on a scale | 1.43 (0.27) | 0.84 (0.27) | 1.57 (0.27)

3. Primary Outcome: Change From Baseline to Week 24 in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (severe disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks
Population: All randomized participants with evaluable HAQ-DI data. Modified Baseline Observation Carried Forward (mBOCF) was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Treatment Period 1 (Weeks 0-52): A loading dose of 2 injections of placebo, followed by maintenance dosing of 1 injection of placebo administered SC Q2W.
  At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  Treatment Period 2 (Weeks 52-100): At Week 52, responders were randomized to receive either 2 injections of 120 mg of LY2127399, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2 or 2 injections of 90 mg of LY2127399, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 327 | 328
units on a scale | -0.26 (0.03) | -0.30 (0.03) | -0.20 (0.03)

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) and 70% (ACR70) Response
Description: ACR Responder Index: Composite of clinical, laboratory, and functional measures of RA. ACR50 Responder: had ≥50% improvement from baseline in both 68 tender joint (TJ) and 66 swollen joint (SJ) counts and ≥50% improvement in at least 3 of 5 criteria: participant's (Pt's) and physician's global assessment of disease activity, HAQ-DI (measured Pts' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of Pt achieving ACR50 response=(number (No.) of ACR50 responders) / (No. of Pts treated) * 100. ACR70 Responder: had ≥70% improvement from baseline in both TJ and SJ counts and ≥70% improvement in at least 3 of same 5 criteria for ACR50. Percentage of Pts achieving ACR70 response= (No. of ACR70 responders) / (No. of Pts treated) * 100. All NR at Week 16 as well as all Pts who discontinued study treatment at any time for any reason were defined as NR starting at that time-point and going forward, including Weeks 24 and 52 endpoints.
Time Frame: Baseline through 24 weeks and 52 weeks
Population: All randomized participants with evaluable ACR50 or ACR70 responder data. If participant's CRP was missing, last post-baseline value was used. If ACR was missing after carrying forward CRP, last post-baseline ACR response was used. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 330 | 332 | 335
percentage of participants
  ACR50 - Week 24 | 10.6 | 11.1 | 10.1
  ACR50 - Week 52 | 4.2 | 3.0 | 4.8
  ACR70 - Week 24 | 3.9 | 3.0 | 3.0
  ACR70 - Week 52 | 1.5 | 1.2 | 1.8

5. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joint Count and C-Reactive Protein Level (DAS28-CRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP [milligrams per liter (mg/L)], and participant's global assessment of disease activity using visual analog scale (VAS) (participant global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*participant global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity and remission is DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable DAS28-CRP data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 328 | 327 | 328
units on a scale
  Week 24 | -1.02 (0.07) | -1.00 (0.07) | -0.78 (0.07)
  Week 52 | -1.07 (0.07) | -1.00 (0.07) | -0.80 (0.07)

6. Secondary Outcome: Percentage of Participants With DAS28-CRP Based European League Against Rheumatism (EULAR) Response
Description: EULAR Responder index based on 28 joint counts categorizes clinical response based on improvement since baseline in DAS28-CRP. DAS28-CRP scores range from 1.0-9.4, where lower scores indicated less disease activity. High disease activity: DAS28-CRP >5.1, low disease activity: DAS28-CRP <3.2, and remission: DAS28-CRP <2.6. Participants are categorized as EULAR responders or NR based on improvement of DAS28-CRP scores from baseline. EULAR DAS28-CRP responder index defines a good (absolute: <3.2 or >1.2 improvement from baseline), moderate (absolute: 3.2-5.1 or 0.6-1.2 improvement from baseline), or no response (absolute: >5.1 or <0.6 improvement from baseline). Percentage of participants with DAS28-CRP based EULAR response =(number of participants with specific response) / (number of participants analyzed in the group) * 100.
Time Frame: Baseline through 24 weeks and 52 weeks
Population: All randomized participants with evaluable EULAR response data. Modified last observation carried forward (mLOCF) was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 328 | 327 | 328
percentage of participants
  Week 24- Good | 17.7 | 16.2 | 14.3
  Week 24 - Moderate | 41.5 | 38.5 | 30.8
  Week 24 - No Response | 40.9 | 45.3 | 54.9
  Week 52 - Good | 18.6 | 14.7 | 15.9
  Week 52 - Moderate | 37.5 | 39.1 | 29.0
  Week 52 - No Response | 43.9 | 46.2 | 55.2

7. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form (SF-36) Health Survey Domain Scores and Summary Scores
Description: SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, 2 component scores (CS), physical CS (PCS) and mental CS (MCS). Domain scores were calculated by summing each item for each domain and transforming scores into a 0-100 scale. Higher scores indicated better health status. If < 50% of the questions within a domain were answered, raw scores were not calculated. PCS score consisted of physical functioning, bodily pain, role-physical, and general health scales. MCS score consisted of social functioning, vitality, mental health, and role-emotional scales. Both PCS and MCS range from 0-100. Higher score indicated better mental or physical health. LS means were calculated using ANCOVA with treatment, region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable SF-36 domain and summary scores. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 320 | 322 | 323
units on a scale
  Physical functioning - Week 24 | 2.70 (0.48) | 3.16 (0.47) | 2.06 (0.47)
  Physical functioning - Week 52 | 2.15 (0.50) | 3.22 (0.49) | 1.82 (0.49)
  Bodily pain - Week 24: number analyzed (Participants) | 319 | 322 | 323
  Bodily pain - Week 24 | 4.07 (0.46) | 4.08 (0.45) | 2.52 (0.45)
  Bodily pain - Week 52: number analyzed (Participants) | 319 | 322 | 323
  Bodily pain - Week 52 | 3.77 (0.47) | 4.48 (0.46) | 2.32 (0.46)
  RL - physical problems - Week 24 | 2.77 (0.46) | 3.64 (0.46) | 1.99 (0.45)
  RL - physical problems - Week 52 | 3.01 (0.47) | 3.79 (0.46) | 1.82 (0.46)
  RL - emotional problems- Week 24: number analyzed (Participants) | 319 | 322 | 323
  RL - emotional problems- Week 24 | 3.20 (0.60) | 4.81 (0.59) | 2.91 (0.59)
  RL - emotional problems- Week 52: number analyzed (Participants) | 319 | 322 | 323
  RL - emotional problems- Week 52 | 2.84 (0.61) | 4.34 (0.59) | 2.56 (0.59)
  GH Perception - Week 24: number analyzed (Participants) | 319 | 322 | 323
  GH Perception - Week 24 | 2.60 (0.41) | 3.72 (0.40) | 2.54 (0.40)
  GH Perception - Week 52: number analyzed (Participants) | 319 | 322 | 323
  GH Perception - Week 52 | 2.89 (0.42) | 3.41 (0.41) | 2.18 (0.41)
  Mental Health - Week 24: number analyzed (Participants) | 319 | 322 | 323
  Mental Health - Week 24 | 3.39 (0.53) | 4.47 (0.53) | 3.28 (0.52)
  Mental Health - Week 52: number analyzed (Participants) | 319 | 322 | 323
  Mental Health - Week 52 | 3.01 (0.55) | 4.37 (0.54) | 3.10 (0.54)
  Social function - Week 24: number analyzed (Participants) | 319 | 322 | 323
  Social function - Week 24 | 3.25 (0.53) | 4.18 (0.52) | 2.79 (0.52)
  Social function - Week 52: number analyzed (Participants) | 319 | 322 | 323
  Social function - Week 52 | 3.04 (0.53) | 3.99 (0.52) | 2.87 (0.52)
  Vitality - Week 24: number analyzed (Participants) | 319 | 322 | 323
  Vitality - Week 24 | 3.43 (0.50) | 4.41 (0.49) | 2.99 (0.48)
  Vitality - Week 52: number analyzed (Participants) | 319 | 322 | 323
  Vitality - Week 52 | 3.10 (0.51) | 3.96 (0.50) | 3.02 (0.49)
  PCS - Week 24: number analyzed (Participants) | 319 | 322 | 323
  PCS - Week 24 | 2.80 (0.43) | 3.08 (0.43) | 1.76 (0.42)
  PCS - Week 52: number analyzed (Participants) | 319 | 322 | 323
  PCS - Week 52 | 2.79 (0.44) | 3.30 (0.43) | 1.55 (0.43)
  MCS - Week 24: number analyzed (Participants) | 319 | 322 | 323
  MCS - Week 24 | 3.34 (0.56) | 4.74 (0.55) | 3.33 (0.55)
  MCS - Week 52: number analyzed (Participants) | 319 | 322 | 323
  MCS - Week 52 | 2.98 (0.57) | 4.27 (0.56) | 3.22 (0.56)

8. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI) Individual Items and Impact Score
Description: The BFI is a brief participant-reported questionnaire for the rapid assessment of fatigue severity and the impact of fatigue on daily functioning in the past 24 hours. The BFI contains 10 items; however, Item 1 is not included in the scoring of the scale as it asks about usual fatigue over the past week with the participant answering 'yes' or 'no'. The remaining 9 items assess fatigue severity (3 items) and impact of fatigue on daily functioning (6 items) using an 11-point numeric scale, with 0=no fatigue and 10=fatigue as bad as you can imagine. The fatigue impact subscale score is the average of the non-missing responses to 6 items: general activity, mood, walking ability, normal work, relations with other people, and enjoyment of life. If more than 3 items within the fatigue impact subscale were not answered by a participant, the subscale is set to missing. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable BFI data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 320 | 322 | 323
units on a scale
  Fatigue-Now - Week 24 | -0.86 (0.14) | -1.12 (0.13) | -0.61 (0.13)
  Fatigue-Now - Week 52 | -0.79 (0.14) | -1.01 (0.13) | -0.56 (0.13)
  Fatigue-Usual - Week 24 | -0.93 (0.13) | -1.06 (0.13) | -0.61 (0.13)
  Fatigue-Usual - Week 52 | -0.91 (0.14) | -0.97 (0.13) | -0.66 (0.13)
  Fatigue-Worst - Week 24 | -0.98 (0.14) | -1.22 (0.14) | -0.71 (0.14)
  Fatigue-Worst - Week 52 | -1.22 (0.15) | -1.19 (0.14) | -0.81 (0.14)
  General Activity - Week 24 | -0.93 (0.14) | -1.09 (0.13) | -0.61 (0.13)
  General Activity - Week 52 | -1.03 (0.14) | -1.07 (0.13) | -0.61 (0.13)
  Mood - Week 24 | -0.67 (0.14) | -1.01 (0.14) | -0.47 (0.14)
  Mood - Week 52 | -0.86 (0.14) | -0.82 (0.14) | -0.53 (0.14)
  Walking Ability - Week 24 | -0.92 (0.15) | -1.02 (0.14) | -0.44 (0.14)
  Walking Ability - Week 52 | -0.88 (0.14) | -0.98 (0.14) | -0.45 (0.14)
  Normal Work - Week 24: number analyzed (Participants) | 320 | 322 | 322
  Normal Work - Week 24 | -0.78 (0.14) | -1.07 (0.14) | -0.48 (0.14)
  Normal Work - Week 52 | -0.88 (0.14) | -1.00 (0.14) | -0.52 (0.14)
  Relations with Other - Week 24: number analyzed (Participants) | 320 | 322 | 322
  Relations with Other - Week 24 | -0.39 (0.14) | -0.64 (0.14) | -0.13 (0.14)
  Relations with Other - Week 52 | -0.47 (0.14) | -0.46 (0.14) | -0.16 (0.14)
  Enjoyment of Life - Week 24: number analyzed (Participants) | 320 | 322 | 322
  Enjoyment of Life - Week 24 | -0.58 (0.15) | -0.82 (0.15) | -0.36 (0.14)
  Enjoyment of Life - Week 52 | -0.66 (0.15) | -0.74 (0.14) | -0.46 (0.14)
  Fatigue Impact Subscale- Week 24 | -0.71 (0.13) | -0.93 (0.13) | -0.42 (0.13)
  Fatigue Impact Subscale- Week 52 | -0.80 (0.13) | -0.83 (0.13) | -0.46 (0.13)

9. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness (Minutes)
Description: The Investigator asks participants about the duration of their morning stiffness (in minutes) in and around the joints and records the duration. The Investigator should ask the participants about duration of morning stiffness on the day prior to the study visit to capture actual symptoms. If morning stiffness duration is longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable morning stiffness data; mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 307 | 319 | 314
minutes
  Week 24: number analyzed (Participants) | 306 | 318 | 313
  Week 24 | -41.2 (5.0) | -32.0 (4.8) | -34.5 (4.9)
  Week 52 | -41.4 (5.2) | -31.2 (5.0) | -37.3 (5.1)

10. Secondary Outcome: Change From Baseline in Brief Pain Inventory Short Form (BPI-SF) Individual Items and Interference Scores
Description: The BPI-SF is a self-reported scale that measures the severity of pain based on the worst pain, least pain, average pain experienced during the past 24-hours and pain based on the pain right now with scores ranging from 0 (no pain) to 10 (pain as severe as you can imagine). Pain interference score is the average of the responses in past 24-hours to 7 items: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life [each item scored from 0 (does not interfere) to 10 (completely interferes)]. If more than 3 items of the Pain Interference Score are not answered by a participant, the score were set to missing. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable BPI-SF scores. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 320 | 322 | 323
units on a scale
  Pain-Worst - Week 24 | -1.1 (0.1) | -1.1 (0.1) | -0.7 (0.1)
  Pain-Worst - Week 52 | -1.1 (0.1) | -1.3 (0.1) | -0.8 (0.1)
  Pain-Least - Week 24 | -0.3 (0.1) | -0.6 (0.1) | -0.1 (0.1)
  Pain-Least - Week 52 | -0.3 (0.1) | -0.6 (0.1) | -0.1 (0.1)
  Pain-Average - Week 24 | -0.8 (0.1) | -0.9 (0.1) | -0.3 (0.1)
  Pain-Average - Week 52 | -0.7 (0.1) | -1.0 (0.1) | -0.3 (0.1)
  Pain-Now - Week 24 | -1.1 (0.1) | -1.2 (0.1) | -0.5 (0.1)
  Pain-Now - Week 52 | -1.0 (0.1) | -1.3 (0.1) | -0.5 (0.1)
  General Activity - Week 24 | -1.0 (0.1) | -1.0 (0.1) | -0.6 (0.1)
  General Activity - Week 52 | -1.0 (0.1) | -1.2 (0.1) | -0.8 (0.1)
  Mood - Week 24 | -0.9 (0.1) | -1.0 (0.1) | -0.6 (0.1)
  Mood - Week 52 | -1.0 (0.1) | -1.1 (0.1) | -0.7 (0.1)
  Walking Ability - Week 24 | -0.9 (0.1) | -1.2 (0.1) | -0.5 (0.1)
  Walking Ability - Week 52 | -0.8 (0.1) | -1.1 (0.1) | -0.6 (0.1)
  Normal Work - Week 24 | -1.0 (0.1) | -1.0 (0.1) | -0.6 (0.1)
  Normal Work - Week 52 | -0.9 (0.1) | -1.1 (0.1) | -0.6 (0.1)
  Relations with Other - Week 24 | -0.5 (0.1) | -0.6 (0.1) | -0.3 (0.1)
  Relations with Other - Week 52 | -0.5 (0.1) | -0.5 (0.1) | -0.3 (0.1)
  Sleep - Week 24 | -1.0 (0.1) | -1.1 (0.1) | -0.4 (0.1)
  Sleep - Week 52 | -0.9 (0.1) | -1.0 (0.1) | -0.5 (0.1)
  Enjoyment of Life - Week 24 | -0.8 (0.1) | -1.2 (0.1) | -0.5 (0.1)
  Enjoyment of Life - Week 52 | -0.9 (0.1) | -1.1 (0.1) | -0.5 (0.1)
  Pain Interference Score - Week 24 | -0.89 (0.12) | -1.02 (0.12) | -0.50 (0.12)
  Pain Interference Score - Week 52 | -0.85 (0.12) | -1.00 (0.12) | -0.58 (0.12)

11. Secondary Outcome: Percentage of Participants With Major Clinical Response (MCR) During 52 Weeks
Time Frame: Baseline through 52 weeks
Population: Zero participants analyzed. Per protocol and statistical analysis plan (SAP) amendments, the major clinical response classification was not collected for analysis.
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Change From Baseline in mTSS Less Than or Equal to (≤) 0
Description: The mTSS quantifies the extent of bone erosions and joint space narrowing for 44 and 42 joints. X-rays of the hands/wrists and feet are scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosions scores (range=0 to 220 for 44 joints) and narrowing scores (range=0 to 168 for 42 joints) were added to obtain the mTSS (range = 0 [normal] to 388 [maximal disease]). Percentage of participants = (number of participants with mTSS ≤0 at Week 24) / (total number of participants analyzed in the group) * 100.
Time Frame: Baseline through 24 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 295 | 304 | 306
percentage of participants | 61.0 | 61.8 | 56.2

13. Secondary Outcome: Change From Baseline to Week 52 in B Cell Subset Counts
Description: B cell subset counts are: cluster designation (CD)19+ B cell counts, Immature/transitional [CD19+immunoglobulin D (IgD)-CD27-], Mature naïve (CD19+IgD+CD27-), Non-switched memory (CD19+IgD+CD27+) and Memory (CD19+IgD-CD27+). A positive or negative change indicated an increase or decrease, respectively in B cell count. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with evaluable B cell subset counts data. mLOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: cells/microliter (cells/µL)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 326 | 333 | 339
cells/microliter (cells/µL)
  CD19+ | -57.1 (4.9) | -60.9 (4.9) | 0.7 (4.8)
  CD19+IgD-CD27-: number analyzed (Participants) | 321 | 330 | 336
  CD19+IgD-CD27- | -3.1 (0.7) | -3.9 (0.7) | 0.2 (0.7)
  CD19+IgD+CD27-: number analyzed (Participants) | 321 | 330 | 336
  CD19+IgD+CD27- | -89.4 (3.3) | -92.4 (3.3) | -3.5 (3.2)
  CD19+IgD+CD27+: number analyzed (Participants) | 321 | 330 | 336
  CD19+IgD+CD27+ | 9.5 (1.0) | 8.9 (1.0) | 1.0 (1.0)
  CD19+IgD-CD27+: number analyzed (Participants) | 321 | 330 | 336
  CD19+IgD-CD27+ | 19.7 (1.9) | 20.6 (1.8) | 3.2 (1.8)

14. Secondary Outcome: Population Pharmacokinetics (PK): Constant Clearance
Description: Population estimate of constant clearance as determined by population PK analysis. A 2-compartment model was used in PK modeling. Constant clearance is the PK parameter which describes the linear elimination of LY2127399 from serum.
Time Frame: Baseline through 52 weeks
Population: All randomized participants who received at least 1 dose of LY2127399 with evaluable LY2127399 PK data.
Measure: Mean (95% Confidence Interval); unit: milliliter per hour (mL/h)
Groups:
- LY2127399: A loading dose of 240 mg (2 injections of 120 mg) of LY2127399 followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 100 weeks or a loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 100 weeks. At Weeks 16 and 52, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 100-week treatment period or 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 100-week treatment period.
Arm/Group | LY2127399
Number analyzed (Participants) | 825
milliliter per hour (mL/h) | 3.60 [3.46 to 3.73]

15. Secondary Outcome: Percentage of Participants Developing Anti-LY2127399 Antibodies
Description: Participants with treatment-emergent anti-drug antibodies (ADA) were participants who had any sample from baseline up to and through Week 24 that was a 4-fold increase (2-dilution increase) in immunogenicity titer over baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20). Percentage of participants with ADA=(number of participants with treatment-emergent ADA) / (number of participants assessed) * 100.
Time Frame: Baseline through 52 weeks
Population: All randomized participants who received at least 1 dose of study drug with an evaluable baseline ADA result and a post-baseline ADA result. Participants missing an evaluable baseline result with all negative post-baseline results were included. Data after Week 16 for Week 16 NR were not included.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 344 | 344 | 347
percentage of participants | 3.8 | 1.5 | 4.9

16. Secondary Outcome: Percentage of Participants With No Structural Progression at Week 52
Description: No structural progression is defined as the change in mTSS from baseline ≤0. The mTSS quantifies the extent of bone erosions and joint space narrowing for 44 and 42 joints. X-rays of the hands/wrists and feet are scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosions scores (range=0 to 220 for 44 joints) and narrowing scores (range=0 to 168 for 42 joints) were added to obtain the mTSS (range=0 [normal] to 388 [maximal disease]). Percentage of participants=(number of participants with mTSS ≤0 at Week 52) / (total number of participants analyzed in the group) * 100.
Time Frame: Baseline through 52 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 295 | 304 | 306
percentage of participants | 55.6 | 57.6 | 53.9

17. Secondary Outcome: Change From Baseline to Week 24 in mTSS
Description: The mTSS quantifies the extent of bone erosions and joint space narrowing for 44 and 42 joints. X-rays of the hands/wrists and feet are scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosions scores (range=0 to 220 for 44 joints) and narrowing scores (range=0 to 168 for 42 joints) were added to obtain the mTSS (range=0 [normal] to 388 [maximal disease]). LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 295 | 304 | 306
units on a scale | 0.63 (0.14) | 0.45 (0.14) | 0.82 (0.14)

18. Secondary Outcome: Change From Baseline in Serum Immunoglobulin (Ig) Levels
Description: Immunoglobulins (Ig), or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Change from baseline serum immunoglobulin G (IgG), immunoglobulin A (IgA), and immunoglobulin M (IgM) levels are reported. A negative change indicated a decrease in Ig levels. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with evaluable serum Ig data. mLOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: grams/liter (g/L)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 342 | 342 | 347
grams/liter (g/L)
  IgA | -0.380 (0.028) | -0.382 (0.028) | -0.009 (0.028)
  IgG | -1.375 (0.096) | -1.235 (0.097) | -0.176 (0.096)
  IgM | -0.235 (0.016) | -0.274 (0.016) | -0.032 (0.016)

19. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score and Bone Erosions Score (Components of mTSS)
Description: as for outcome 17
Time Frame: Baseline, 24 weeks and 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 295 | 304 | 306
units on a scale
  Joint Space Narrowing - Week 24 | 0.22 (0.09) | 0.19 (0.09) | 0.34 (0.09)
  Joint Space Narrowing - Week 52 | 0.56 (0.16) | 0.35 (0.16) | 0.61 (0.16)
  Bone Erosions - Week 24 | 0.40 (0.09) | 0.26 (0.08) | 0.48 (0.08)
  Bone Erosions - Week 52 | 0.86 (0.17) | 0.49 (0.17) | 0.96 (0.17)

20. Secondary Outcome: American College of Rheumatology Percent Improvement (ACR-N)
Description: ACR-N is a continuous measure of clinical, laboratory, and functional outcomes in RA that characterizes percentage (%) of improvement in disease activity from baseline based on ACR core set. This index was calculated as minimum of either a) % change in TJ count, b) % change in SJ count, or c) the median % change of remaining 5 ACR core criteria: If ≥3 components of the 5 ACR core criteria were missing, then c) was set to missing; if any of 3 components a), b), or c) were missing, then ACR-N was set to missing. Percentage of improvement was truncated to range of -100 to 100 to minimize impact of outliers (greater values indicate greater % improvement) and negative scores indicate a decline. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline DAS28-CRP as a covariate.
Time Frame: Baseline through 24 weeks and 52 weeks
Population: All randomized participants with evaluable ACR-N data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: percentage of improvement
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 326 | 327
percentage of improvement
  Week 24 | 2.0 (2.5) | 2.1 (2.5) | -6.9 (2.5)
  Week 52 | 2.9 (2.5) | 0.3 (2.5) | -7.3 (2.5)

21. Secondary Outcome: Change From Baseline in Tender Joint Count (68 Joint Count)
Description: Tender joint count is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable tender joint count data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 329 | 334
joint counts
  Week 24 | -7.41 (0.72) | -7.88 (0.72) | -6.40 (0.72)
  Week 52 | -7.88 (0.73) | -8.09 (0.73) | -5.72 (0.73)

22. Secondary Outcome: Change From Baseline in Swollen Joint Count (66 Joint Count)
Description: Swollen joint count is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable swollen joint count data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 329 | 334
joint counts
  Week 24 | -5.38 (0.49) | -5.64 (0.49) | -4.67 (0.49)
  Week 52 | -6.10 (0.49) | -5.53 (0.49) | -4.61 (0.49)

23. Secondary Outcome: Change From Baseline in Participant's Assessment of Pain [Visual Analog Scale (VAS)]
Description: Participant's assessment of their current arthritis pain using VAS ranged from 0 millimeters (mm) (no pain) to 100 mm (worst possible pain). A decrease in pain score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable participant's assessment of pain data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 327 | 328
units on a scale
  Week 24 | -13.6 (1.2) | -14.6 (1.2) | -9.0 (1.2)
  Week 52 | -13.2 (1.2) | -14.6 (1.2) | -8.7 (1.2)

24. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity (VAS)
Description: Participant's assessment of their current arthritis disease activity using VAS ranged from 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). A decrease in disease activity score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable participant's global assessment of disease activity data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 327 | 328
mm
  Week 24 | -13.2 (1.2) | -15.1 (1.2) | -11.0 (1.2)
  Week 52 | -13.1 (1.2) | -15.2 (1.2) | -10.8 (1.2)

25. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity (VAS)
Description: Physician's assessment of the participant's current arthritis disease activity using VAS ranged from 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). A decrease in disease activity score indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable physician's global assessment of disease activity data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 321 | 315 | 314
mm
  Week 24 | -20.7 (1.3) | -22.0 (1.3) | -17.2 (1.3)
  Week 52 | -20.4 (1.3) | -20.6 (1.3) | -17.8 (1.3)

26. Secondary Outcome: Change From Baseline to Week 52 in HAQ-DI
Description: as for outcome 3
Time Frame: Baseline, 52 weeks
Population: All randomized participants with evaluable HAQ-DI data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 327 | 328
units on a scale | -0.24 (0.03) | -0.30 (0.03) | -0.18 (0.03)

27. Secondary Outcome: Change From Baseline to Week 52 in Absolute B Cell Counts
Description: Cell-surface marker cluster designation (CD) 3 negative, CD20 positive (CD3-CD20+) defines total mature B cells. B-lymphocyte antigen CD20 is an activated-glycosylated phosphoprotein expressed on the surface of all mature B cells. A positive or negative change indicated an increase or decrease, respectively in B cell count. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 52 weeks
Population: All randomized participants with evaluable CD3-CD20+ B cell counts. mLOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: cells/microliter (cells/µL)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 343 | 344 | 348
cells/microliter (cells/µL) | -56.5 (4.5) | -58.6 (4.5) | -6.8 (4.5)

28. Secondary Outcome: Percentage of Participants With ACR20 at Week 52
Description: ACR Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis (RA). ACR20 Responder: had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, HAQ-DI (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and CRP. Percentage of participants achieving ACR20 response=(number of ACR20 responders) /( number of participants treated) * 100. All NR at Week 16 as well as all participants who discontinued study treatment at any time for any reason were defined as NR starting at that time-point and going forward, including Week 52 endpoint.
Time Frame: Baseline through 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 330 | 332 | 335
percentage of participants | 7.9 | 9.6 | 10.7

29. Secondary Outcome: Time to ACR20 Response
Description: ACR Responder Index: Composite of clinical, laboratory, and functional measures of rheumatoid arthritis (RA). ACR20 Responder: had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, HAQ-DI (which measured participants' perceived degree of difficulty performing daily activities), joint pain, and CRP. The Kaplan-Meier was used to estimate time to ACR20 response over the Treatment Period (52 weeks). Time to ACR20 response = (Date of the first post-baseline visit during the Treatment Period meeting ACR20 response criteria - Date of first injection of study treatment + 1) / 7. Week 16 NR are counted as responders if they responded prior to Week 16. Otherwise, they are censored at the date of the Week 16 injection. All participants ongoing at Week 52 and had not yet responded are censored at the date of the Week 52 visit.
Time Frame: Baseline through 52 weeks
Population: All randomized participants with evaluable ACR20 responder data. The number of participants censored are 128 (120 mg LY2127399), 123 (90 mg LY2127399) and 162 (placebo).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 327 | 327 | 329
weeks | 16.1 [12.1 to 16.4] | 16.1 [12.3 to 20.0] | 20.1 [16.4 to 24.7]

30. Secondary Outcome: Change From Baseline in CRP
Description: CRP is an indicator of inflammation. A negative change indicated an improvement in the participant's condition. LS means were calculated using ANCOVA with treatment and region as fixed factors and baseline as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks
Population: All randomized participants with evaluable CRP data. mBOCF was used to impute missing post-baseline values. Data after Week 16 for Week 16 NR were not included.
Measure: Least Squares Mean (Standard Error); unit: milligrams/liter (mg/L)
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 329 | 328 | 334
milligrams/liter (mg/L)
  Week 24 | -3.30 (0.83) | -2.03 (0.84) | -0.54 (0.83)
  Week 52 | -1.72 (0.96) | -2.04 (0.97) | -0.40 (0.96)

31. Other Pre Specified Outcome: Number of Participants Who Died During Post-Treatment Follow-Up Period
Time Frame: Discontinuation from study treatment up to 48 weeks during follow-up period
Population: All randomized participants who received at least 1 dose of study drug and entered post-treatment follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | 120 mg LY2127399 | 90 mg LY2127399 | Placebo
Number analyzed (Participants) | 293 | 303 | 307
Participants | 0 | 1 | 2

ADVERSE EVENTS:
Groups:
- LY 120 mg Q4W, Randomized Treatment Period 1: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 52 weeks during Treatment Period 1. At Week 16, responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 52-week Treatment Period 1. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  The Randomized Treatment Period 1 was defined as the time all data was collected during the Treatment Period 1, excluding the data collected after the date of the Week 16 injection for the Week 16 NR.
- LY 90 mg Q2W, Randomized Treatment Period 1: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, responders received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 1.
  The Randomized Treatment Period 1 was defined as the time all data was collected during the Treatment Period 1, excluding the data collected after the date of the Week 16 injection for the Week 16 NR.
- Placebo, Randomized Treatment Period 1: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  The Randomized Treatment Period 1 was defined as the time all data was collected during the Treatment Period 1, excluding the data collected after the date of the Week 16 injection for the Week 16 NR.
- LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Rescue Period: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 16 weeks during Treatment Period 1. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the Treatment Period 1 for Week 16 NR.
- LY 90 mg Q2W, Rescue Period: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 16 weeks during Treatment Period 1.
  At Week 16, NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the Treatment Period 1 for Week 16 NR.
- Placebo to LY 90 mg Q2W (Week 16), Rescue Period: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 16 weeks during Treatment Period 1.
  At Week 16, NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  The Rescue Treatment Period was defined as all data collected after the date of the Week 16 injection during the Treatment Period 1 for Week 16 NR.
- LY 120 mg Q4W, Treatment Period 2: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 52 weeks during Treatment Period 1. At Week 16, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 52-week Treatment Period 1. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 52, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2.
  Treatment Period 2 was defined as all data collected from Week 52 to Week 100 during non-blinded Treatment Period 2.
- LY 90 mg Q2W, Treatment Period 2: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, both Week 16 responders and NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 1.
  At Week 52, both Week 16 responders and NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
  Treatment Period 2 was defined as all data collected from Week 52 to Week 100 during non-blinded Treatment Period 2.
- Placebo to LY 120 mg Q4W (Week 52), Treatment Period 2: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, Week 16 responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  At Week 52, Week 16 responders were randomized to receive 2 injections of 120 mg of LY2127399, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2
  Treatment Period 2 was defined as all data collected from Week 52 to Week 100 during non-blinded Treatment Period 2.
- Placebo to LY 90 mg Q2W (Week 52), Treatment Period 2: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, Week 16 responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  At Week 52, Week 16 responders were randomized to receive 2 injections of 90 mg of LY2127399, followed by 90 mg of LY2127399 Q4W for the rest of the Treatment Period 2
  Treatment Period 2 was defined as all data collected from Week 52 to Week 100 during non-blinded Treatment Period 2.
- LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Treatment Period 2: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 16 weeks during Treatment Period 1. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, Week 16 NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  During non-blinded Treatment Period 2, Week 16 NR received 1 injection of 90 mg of LY2127399.
  Treatment Period 2 was defined as all data collected from Week 52 to Week 100 during non-blinded Treatment Period 2.
- Placebo to LY 90 mg Q2W (Week 16), Treatment Period 2: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 16 weeks during Treatment Period 1.
  At Week 16, Week 16 NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  During non-blinded Treatment Period 2, Week 16 NR received 1 injection of 90 mg of LY2127399.
  Treatment Period 2 was defined as all data collected from Week 52 to Week 100 during non-blinded Treatment Period 2.
- LY 120 mg Q4W, Follow-up Period: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 52 weeks during Treatment Period 1. At Week 16, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the 52-week Treatment Period 1. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 52, Week 16 responders received 1 injection of 120 mg of LY2127399 and 1 injection of placebo, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2.
  The Post-Treatment Follow-Up Period started after Week 100 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- LY 90 mg Q2W, Follow-up Period: A loading dose of 180 mg of LY2127399 (2 injections of 90 mg) followed by maintenance dosing of 90 mg of LY2127399 administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, both Week 16 responders and NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 1.
  At Week 52, both Week 16 responders and NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the Treatment Period 2.
  The Post-Treatment Follow-Up Period started after Week 100 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo to LY 120 mg Q4W (Week 52), Follow-up Period: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, Week 16 responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  At Week 52, Week 16 responders were randomized to receive 2 injections of 120 mg of LY2127399, followed by 120 mg of LY2127399 Q4W for the rest of the Treatment Period 2
  The Post-Treatment Follow-Up Period started after Week 100 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo to LY 90 mg Q2W (Week 52), Follow-up Period: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, Week 16 responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  At Week 52, Week 16 responders were randomized to receive 2 injections of 90 mg of LY2127399, followed by 90 mg of LY2127399 Q4W for the rest of the Treatment Period 2
  The Post-Treatment Follow-Up Period started after Week 100 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period: A loading dose of 240 mg of LY2127399 (2 injections of 120 mg) followed by maintenance dosing of 120 mg of LY2127399 administered SC Q4W for 16 weeks during Treatment Period 1. For blinding purposes, participants alternated injections of LY2127399 and injections of placebo Q2W.
  At Week 16, Week 16 NR received 1 injection of 90 mg of LY2127399 and 1 injection of placebo, followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  During non-blinded Treatment Period 2, Week 16 NR received 1 injection of 90 mg of LY2127399.
  The Post-Treatment Follow-Up Period started after Week 100 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo to LY 90 mg Q2W (Week 16), Follow-up Period: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 16 weeks during Treatment Period 1.
  At Week 16, Week 16 NR received a loading dose of 180 mg of LY2127399 (2 injections of 90 mg), followed by 90 mg of LY2127399 Q2W for the rest of the 52-week Treatment Period 1.
  During non-blinded Treatment Period 2, Week 16 NR received 1 injection of 90 mg of LY2127399.
  The Post-Treatment Follow-Up Period started after Week 100 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
- Placebo, Follow-up Period: A loading dose of 2 injections of placebo followed by maintenance dosing of placebo administered SC Q2W for 52 weeks during Treatment Period 1. At Week 16, responders received 2 injections of placebo, followed by 1 injection of placebo Q2W for the rest of the Treatment Period 1.
  The Post-Treatment Follow-Up Period started after Week 52 or the early discontinuation visit and lasted up to 48 weeks following the last injection of study treatment.
Arm/Group | LY 120 mg Q4W, Randomized Treatment Period 1 | LY 90 mg Q2W, Randomized Treatment Period 1 | Placebo, Randomized Treatment Period 1 | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Rescue Period | LY 90 mg Q2W, Rescue Period | Placebo to LY 90 mg Q2W (Week 16), Rescue Period | LY 120 mg Q4W, Treatment Period 2 | LY 90 mg Q2W, Treatment Period 2 | Placebo to LY 120 mg Q4W (Week 52), Treatment Period 2 | Placebo to LY 90 mg Q2W (Week 52), Treatment Period 2 | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Treatment Period 2 | Placebo to LY 90 mg Q2W (Week 16), Treatment Period 2 | LY 120 mg Q4W, Follow-up Period | LY 90 mg Q2W, Follow-up Period | Placebo to LY 120 mg Q4W (Week 52), Follow-up Period | Placebo to LY 90 mg Q2W (Week 52), Follow-up Period | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period | Placebo to LY 90 mg Q2W (Week 16), Follow-up Period | Placebo, Follow-up Period
Serious Adverse Events (participants affected / at risk) | 19/345 | 17/345 | 17/348 | 3/58 | 3/62 | 2/90 | 1/57 | 1/73 | 2/27 | 1/31 | 0/13 | 0/22 | 9/241 | 14/303 | 1/27 | 1/27 | 5/52 | 4/85 | 14/168
Other Adverse Events (participants affected / at risk) | 137/345 | 117/345 | 129/348 | 22/58 | 25/62 | 20/90 | 22/57 | 20/73 | 7/27 | 4/31 | 7/13 | 9/22 | 43/241 | 39/303 | 6/27 | 9/27 | 10/52 | 10/85 | 26/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY 120 mg Q4W, Randomized Treatment Period 1 (N=345) | LY 90 mg Q2W, Randomized Treatment Period 1 (N=345) | Placebo, Randomized Treatment Period 1 (N=348) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Rescue Period (N=58) | LY 90 mg Q2W, Rescue Period (N=62) | Placebo to LY 90 mg Q2W (Week 16), Rescue Period (N=90) | LY 120 mg Q4W, Treatment Period 2 (N=57) | LY 90 mg Q2W, Treatment Period 2 (N=73) | Placebo to LY 120 mg Q4W (Week 52), Treatment Period 2 (N=27) | Placebo to LY 90 mg Q2W (Week 52), Treatment Period 2 (N=31) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Treatment Period 2 (N=13) | Placebo to LY 90 mg Q2W (Week 16), Treatment Period 2 (N=22) | LY 120 mg Q4W, Follow-up Period (N=241) | LY 90 mg Q2W, Follow-up Period (N=303) | Placebo to LY 120 mg Q4W (Week 52), Follow-up Period (N=27) | Placebo to LY 90 mg Q2W (Week 52), Follow-up Period (N=27) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period (N=52) | Placebo to LY 90 mg Q2W (Week 16), Follow-up Period (N=85) | Placebo, Follow-up Period (N=168)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/294 (0) | 1/289 (1) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/294 (0) | 1/289 (1) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/294 (1) | 0/289 (0) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/294 (0) | 0/289 (0) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 1/255 (1) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/294 (0) | 0/289 (0) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 1/255 (1) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/294 (1) | 0/289 (0) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY 120 mg Q4W, Randomized Treatment Period 1 (N=345) | LY 90 mg Q2W, Randomized Treatment Period 1 (N=345) | Placebo, Randomized Treatment Period 1 (N=348) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Rescue Period (N=58) | LY 90 mg Q2W, Rescue Period (N=62) | Placebo to LY 90 mg Q2W (Week 16), Rescue Period (N=90) | LY 120 mg Q4W, Treatment Period 2 (N=57) | LY 90 mg Q2W, Treatment Period 2 (N=73) | Placebo to LY 120 mg Q4W (Week 52), Treatment Period 2 (N=27) | Placebo to LY 90 mg Q2W (Week 52), Treatment Period 2 (N=31) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Treatment Period 2 (N=13) | Placebo to LY 90 mg Q2W (Week 16), Treatment Period 2 (N=22) | LY 120 mg Q4W, Follow-up Period (N=241) | LY 90 mg Q2W, Follow-up Period (N=303) | Placebo to LY 120 mg Q4W (Week 52), Follow-up Period (N=27) | Placebo to LY 90 mg Q2W (Week 52), Follow-up Period (N=27) | LY 120 mg Q4W to LY 90 mg Q2W (Week 16), Follow-up Period (N=52) | Placebo to LY 90 mg Q2W (Week 16), Follow-up Period (N=85) | Placebo, Follow-up Period (N=168)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 6 (6) | 11 (11) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 9 (9) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (11) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 4 (5) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 8 (8) | 8 (8) | 11 (11) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 20 (25) | 15 (22) | 25 (34) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 7 (9) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 5 (5)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 18 (21) | 20 (21) | 18 (20) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (12) | 6 (8) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0/294 (0) | 0/289 (0) | 0/291 (0) | 1/44 (1) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 9 (10) | 7 (7) | 2 (8) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12 (14) | 19 (20) | 15 (18) | 3 (3) | 5 (5) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/294 (0) | 0/289 (0) | 0/291 (0) | 0/44 (0) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 1/24 (1) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/294 (1) | 1/289 (1) | 0/291 (0) | 1/44 (1) | 0/57 (0) | 0/69 (0) | 1/51 (1) | 1/62 (1) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (10) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/51 (0) | 1/56 (1) | 0/57 (0) | 0/14 (0) | 1/5 (1) | 0/21 (0) | 0/6 (0) | 0/11 (0) | 0/5 (0) | 0/4 (0) | 0/4 (0) | 0/3 (0) | 0/30 (0) | 1/48 (1) | 0/5 (0) | 0/3 (0) | 0/12 (0) | 0/19 (0) | 0/22 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0/294 (0) | 0/289 (0) | 0/291 (0) | 1/44 (1) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1/294 (1) | 0/289 (0) | 0/291 (0) | 1/44 (1) | 0/57 (0) | 0/69 (0) | 0/51 (0) | 0/62 (0) | 0/22 (0) | 0/27 (0) | 0/9 (0) | 0/19 (0) | 0/211 (0) | 0/255 (0) | 0/22 (0) | 0/24 (0) | 0/40 (0) | 0/66 (0) | 0/146 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 12 (13) | 3 (3) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study has been terminated not based on safety concerns, but due to insufficient efficacy. Early termination led to lower than expected enrollment and was responsible for the large number of discontinuation reason as Sponsor Decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days